CLINICAL TRIAL: NCT06800456
Title: The Role of Cyberchondria Severity in the Relationship Between HPV Awareness and Vaccination Attitudes in Adult Women
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Merve Coskun, Assistant Professor, Acibadem University
Other Study IDs: 2024-7-268
Record Dates: First submitted 2024-07-17; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Human Papillomavirus Infection; HPV Vaccines; Cyberchondria; Awareness; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Papillomavirus Infections; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human papillomavirus (HPV) is a prevalent sexually transmitted infection linked to nearly all cases (99%) of cervical cancer. Prophylactic HPV vaccination is effective in preventing these cancers, complemented by HPV screening and treatment of precancerous lesions. The World Health Organization (WHO) aims to eliminate cervical cancer by 2030 through focused efforts on vaccination, diagnosis, and treatment.

Primary prevention strategies include reducing sexual risk factors and administering prophylactic vaccines. Despite awareness of HPV testing, many women lack understanding of its importance and fail to follow through with screenings and necessary treatments. Overall societal awareness of HPV remains inadequate.

Studies reveal disparities in HPV vaccine awareness: while 60.7% of women have heard of the vaccine, only 1% have received it. Awareness varies widely across regions, with Turkey reporting rates from 3.8% to 57%, and vaccine awareness ranging from 2.2% to 74.7% (Özdemir et al., 2020). In the UK, concerns over potential negative results lead many women to defer HPV testing.

Health anxiety, defined as interpreting minor symptoms as serious health issues, drives individuals to seek excessive online health information, a phenomenon known as cyberchondria. Studies link cyberchondria with heightened health anxiety, exacerbated by prolonged internet searches.

Barriers to HPV screening and vaccination include fear of side effects, lack of information, cost concerns, and anxiety over potential outcomes. While women testing positive for HPV show higher levels of cyberchondria, no direct correlation has been established between cyberchondria severity and HPV awareness or vaccination attitudes in adult women.

This summary encapsulates the key findings and insights from the referenced studies on HPV, vaccination, and health anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-49 years old
* At least elementary school education

Exclusion Criteria:

* Individuals diagnosed with psychiatric disorders
* Women who are HPV (Human Papilloma Virus) positive
* Any condition that would hinder communication (e.g., language barrier)

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: The study includes women aged 18-49 years, who have completed at least elementary school education. The study aims to explore awareness and concern levels regarding HPV (Human Papilloma Virus) among women within the specified age range and educational background.
Sampling Method: Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Introduction Information Forum | Upon presentation to the clinic
  This form, prepared by researchers in accordance with the literature, includes general questions about women's sociodemographic characteristics, reproductive health, and health-seeking behaviors. The form consists of a total of 32 questions
Human Papilloma Virus Awareness and Concern Scale for Women (Women HPV-ACS) | Upon presentation to the clinic
  Developed by Esencan et al. (2023), this scale aims to measure awareness and concern levels related to Human Papilloma Virus (HPV). The scale comprises 19 items organized into three subscales. Scores range from 0 to 76, with higher scores indicating greater awareness of HPV. The subscales include: Concerns about health (items 7, 8, 9, 10, 11, 12, 13, 14), Concerns about social exclusion (items 15, 16, 17, 18, 19), and Awareness (items 1, 2, 3, 4, 5, 6). Responses are rated on a 5-point Likert scale ranging from 0 (Definitely disagree) to 4 (Definitely agree). The Cronbach's Alpha reliability coefficient for the scale is 0.905 (Esencan et al., 2023)
Cyberchondria Severity Scale Short Form (CSS-SF) | Upon presentation to the clinic
  Developed by McElroy and Shevlin in 2019 and validated by Yam et al. (2023), the CSS-SF consists of 12 items assessing the severity of online symptom searching behaviors related to health concerns. The scale includes four subscales: Excessiveness, Distress, Reassurance-seeking, and Compulsion. Responses are rated on a 5-point Likert scale ranging from 1 (Never) to 5 (Always). Total scores range from 5 to 60, with higher scores indicating greater severity of cyberchondria. The total Cronbach's Alpha coefficient for the scale is 0.89, with subscale Cronbach's Alpha values ranging as follows: 0.83, 0.79, 0.70, 0.80 (Yam et al., 2023).
  These descriptions outline the key measures used in the study to assess awareness and concern levels regarding HPV and severity of cyberchondria among women.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Coşkun, phd, Principal Investigator — Acibadem University; İrem Nur Özdemir, phd, Principal Investigator — Bakirköy Dr.Sadi Konuk Trainng and Research Hospital
Locations (1):
- Güzin Ünlü Suvari, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agrawal V, Khulbe Y, Singh A, Kar SK. The digital health dilemma: Exploring cyberchondria, well-being, and smartphone addiction in medical and non-medical undergraduates. Indian J Psychiatry. 2024 Mar;66(3):256-262. doi: 10.4103/indianjpsychiatry.indianjpsychiatry_570_23. Epub 2024 Mar 18. PMID 39100122
- [Background] Barke A, Bleichhardt G, Rief W, Doering BK. The Cyberchondria Severity Scale (CSS): German Validation and Development of a Short Form. Int J Behav Med. 2016 Oct;23(5):595-605. doi: 10.1007/s12529-016-9549-8. PMID 26931780
- [Background] Baumgartner SE, Hartmann T. The role of health anxiety in online health information search. Cyberpsychol Behav Soc Netw. 2011 Oct;14(10):613-8. doi: 10.1089/cyber.2010.0425. Epub 2011 May 6. PMID 21548797
- [Background] Dany M, Chidiac A, Nassar AH. Human papillomavirus vaccination: assessing knowledge, attitudes, and intentions of college female students in Lebanon, a developing country. Vaccine. 2015 Feb 18;33(8):1001-7. doi: 10.1016/j.vaccine.2015.01.009. Epub 2015 Jan 15. PMID 25597945
- [Background] Eskisu M, Cam Z, Boysan M. Health-Related Cognitions and Metacognitions Indirectly Contribute to the Relationships Between Impulsivity, Fear of COVID-19, and Cyberchondria. J Ration Emot Cogn Behav Ther. 2023 Jan 9:1-23. doi: 10.1007/s10942-022-00495-7. Online ahead of print. PMID 36687465
- [Background] Guvenc G, Seven M, Akyuz A. Health Belief Model Scale for Human Papilloma Virus and its Vaccination: Adaptation and Psychometric Testing. J Pediatr Adolesc Gynecol. 2016 Jun;29(3):252-8. doi: 10.1016/j.jpag.2015.09.007. Epub 2015 Sep 26. PMID 26409648
- [Background] Hendry M, Pasterfield D, Lewis R, Clements A, Damery S, Neal RD, Adke R, Weller D, Campbell C, Patnick J, Sasieni P, Hurt C, Wilson S, Wilkinson C. Are women ready for the new cervical screening protocol in England? A systematic review and qualitative synthesis of views about human papillomavirus testing. Br J Cancer. 2012 Jul 10;107(2):243-54. doi: 10.1038/bjc.2012.256. Epub 2012 Jun 14. PMID 22699825
- [Background] Mousavi, T., Rezapour, M., Moosazadeh, M., Ghaffari, N., & Nazari, Z. (2023). The relationship between the level of knowledge about human papillomavirus and the level of anxiety and sexual satisfaction in women with a positive HPV test. Journal of Mazandaran University of Medical Sciences, 33(2), 329-334.
- [Background] Norr AM, Allan NP, Boffa JW, Raines AM, Schmidt NB. Validation of the Cyberchondria Severity Scale (CSS): replication and extension with bifactor modeling. J Anxiety Disord. 2015 Apr;31:58-64. doi: 10.1016/j.janxdis.2015.02.001. Epub 2015 Feb 14. PMID 25734759
- [Background] Ozdemir S, Akkaya R, Karasahin KE. Analysis of community-based studies related with knowledge, awareness, attitude, and behaviors towards HPV and HPV vaccine published in Turkey: A systematic review. J Turk Ger Gynecol Assoc. 2020 Jun 8;21(2):111-123. doi: 10.4274/jtgga.galenos.2019.2019.0071. Epub 2019 Aug 9. PMID 31397145
- [Background] Patel H, Moss EL, Sherman SM. HPV primary cervical screening in England: Women's awareness and attitudes. Psychooncology. 2018 Jun;27(6):1559-1564. doi: 10.1002/pon.4694. Epub 2018 Apr 16. PMID 29521462
- [Background] Starcevic V, Schimmenti A, Billieux J, Berle D. Cyberchondria in the time of the COVID-19 pandemic. Hum Behav Emerg Technol. 2021 Jan;3(1):53-62. doi: 10.1002/hbe2.233. Epub 2020 Nov 23. PMID 33363277
- [Background] Turhan Cakir A. Cyberchondria levels in women with human papilloma virus. J Obstet Gynaecol Res. 2022 Oct;48(10):2610-2614. doi: 10.1111/jog.15354. Epub 2022 Jul 8. PMID 35801694
- [Background] World Health Organization. (2021). WHO guideline for screening and treatment of cervical precancer lesions for cervical cancer prevention, second edition. Geneva: World Health Organization. Retrieved from https://www.who.int/publications/i/item/9789240014107
- [Background] Yılmaz, B., Hat, B. N., Yürekli, Y., & Oskay, Ü. (2021). Genç erişkinlerin human papilloma virüs (HPV) ve hpv aşısına ilişkin bilgi ve görüşleri: Kesitsel bir çalışma. KOU Sag Bil Derg, 7(2), 138-148.
- [Derived] Coskun M, Unlu Suvari G, Ozdemir IN. Role of cyberchondria severity in the relationship between HPV awareness and vaccination status among adult women. BMC Public Health. 2025 Dec 17. doi: 10.1186/s12889-025-25938-5. Online ahead of print. PMID 41408614